CLINICAL TRIAL: NCT06441357
Title: Differentiating the Invasiveness of Lung Adenocarcinoma by Dual Energy CT Using Extracellular Volume Measured in Delay Phase
Brief Title: Differentiating the Invasiveness of Lung Adenocarcinoma by Dual Energy CT Parameter
Status: Recruiting | Type: Observational
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TDFS20240328
Record Dates: First submitted 2024-05-28; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Adenocarcinoma of Lung
Keywords: ECV, invasion, lung adenocarcinoma, DECT
MeSH Terms: conditions — Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with preinvasive lung adenocarcinomas: preinvasive lung adenocarcinomas include atypical adenomatous hyperplasia (AAH), adenocarcinoma in situ (AIS) and minimally invasive adenocarcinoma (MIA)
- Patients with invasive lung adenocarcinomas: invasive adenocarcinoma(IAC)

SUMMARY:
The core purpose of this study is to investigate whether the extracellular volume (ECV) fraction measured in delay phase by dual energy computed tomography (DECT) can distinguish precancerous lesions from early-stage lung adenocarcinomas, which could assist clinical decision making for surgery operation indication and strategy.

DETAILED DESCRIPTION:
Although progression of lung adenocarcinoma (LUAD) depends on driver mutations, it is also affected by tumor microenvironment (TME), including vessels, immune cells and extracellular matrix (ECM). As major constituent of TME, ECM mediates interactions between cancer cells and stromal cells, promotes angiogenesis, epithelial-mesenchymal transition, causes metastasis and resistance to immune therapy. Along with the progression of LUAD histologic stages, from atypical adenomatous hyperplasia (AAH) and adenocarcinoma in situ (AIS) to minimally invasive adenocarcinoma (MIA), and finally to invasive adenocarcinoma (IA), the composition of the ECM changes a lot, which has some characterizations same as interstitial pulmonary fibrosis. Hence, identifying the pathological ECM status may help differentiating the invasiveness of lung adenocarcinomas.

Based on the theory that in delay phase, the contrast medium is evenly distributed in the intravascular and extravascular-extracellular spaces and not entering the cell, extracellular volume (ECV) fraction is considered as a potential quantitative imaging parameter for ECM. It has been confirmed that ECV fraction is highly consistent with pathological fibrosis in cardiac and hepatic diseases. In other lesions with fibrosis such as pancreatic and thymic epithelial tumors, ECV fraction also has positive effects in malignancy prediction. It has been verified that ECV fraction is capable of differentiating lung cancer with benign lung lesions and classifying lung cancers into three subtypes. However, there has yet no study testified it as an invasion predictor.

The core purpose of this study is to investigate whether ECV fraction can distinguish precancerous lesions from early-stage lung adenocarcinomas and compare it with other confirmed radiological features in prediction performance, which is clinically meaningful regarding optimal treatment selection and avoidance of unnecessary surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years old with pulmonary nodules (diameter≤3 cm).
* pathologically confirmed as lung adenocarcinoma.
* without history of other malignancies.
* accurate hematocrit within 1 week before contrast enhanced dual energy CT examination.

Exclusion Criteria:

* with a history of allergy to iodine contrast agents and other reasons who are unable to complete the examination.
* without histopathology of invasion stage, such as AAH, AIS, MIA and IAC.
* history of chemotherapy, radiotherapy, or other anti-tumor therapy before contrast enhanced dual energy CT.
* poor image quality.
* contrast enhanced dual energy CT scans ≥ 4 weeks before surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pulmonary nodules who intend to have contrast enhanced CT in Tangdu hospital.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Acquire DECT parameters in patients with pulmonary nodules. | 2 years
  Including iodine concentration (IC) in delay phase, normalized IC (NIC), effective atomic number (Zeff), and CT attenuation values of nodules from virtual monochromatic images (VMIs) (energy range from 40 to 150 keV, 10keV as interval).

OTHER OUTCOMES:
Acquire relative radiological features. | 2 years
  Including consolidation tumor ratio (CTR), nodule's maximum diameter, spiculation, lobulation, fibrosis, distortion or cut-off of vessels and bronchi.

CONTACTS AND LOCATIONS:
Overall Officials: Cui Guangbin, Study Chair — ang-Du Hospital
Locations (1):
- Tangdu Hospital, Xi'an, Shaanxi, China